CLINICAL TRIAL: NCT02326506
Title: Evaluation of Drainable Volume Measurements and Their Usage for Predicting Optimal Cardiac Support in Patients Supported by Veno-arterial Extracorporeal Life Support
Brief Title: Evaluation of Drainable Volume Measurements During VA-ELS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL49011.000.14
Record Dates: First submitted 2014-10-08; First posted 2014-12-29 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Heart Arrest
Keywords: Extracorporeal Membrane Oxygenation; Cardiopulmonary Bypass
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pump speed variation (Experimental): VA-ELS pump speed variations
  Interventions: Device: VA-ELS pump speed variations

INTERVENTIONS:
Device: VA-ELS pump speed variations — Small variations in the pump speed of the veno-arterial extracorporeal life support (VA-ELS) pump

SUMMARY:
Veno-arterial extracorporeal life support (VA-ELS) is used to support patients with acute cardiac failure. In that context, sufficient drainable venous volume is crucial for reliable and adequate support. To date, no reliable measurement method exists to monitor drainable volume adequately. Furthermore, it is still unresolved how to diagnose adequate cardiac recovery.

Previous (pre)clinical studies showed that the calculation of the dynamic filling index may provide a valuable parameter to monitor the drainable volume in patients supported by VAELS. In addition, a case report showed that measurement of the dynamic filling index could successfully be used to estimate cardiac recovery in a single patient supported by VA-ELS in the ICU.

This study will assess the dynamic filling index as a representation for drainable volume and cardiac recovery using standard recorded perfusion data in patients supported by VA-ELS

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the relative(s) or legal representative(s)
* Supported by VA-ELS at the ICU
* >18 years

Exclusion Criteria:

- Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
TEE results | participants will be followed for the duration of the VA-ELS support, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W. Weerwind, Dr., Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Hospital, Maastricht, Netherlands

REFERENCES:
- [Background] Simons AP, Reesink KD, Lance MD, van der Nagel T, van der Veen FH, Weerwind PW, Maessen JG. Reserve-driven flow control for extracorporeal life support: proof of principle. Perfusion. 2010 Jan;25(1):25-9. doi: 10.1177/0267659109360284. Epub 2010 Jan 29. PMID 20118166
- [Background] Simons AP, Reesink KD, Lance MD, van der Veen FH, de Jong DS, Weerwind PW, Maessen JG. Dynamic filling index: a novel parameter to monitor circulatory filling during minimized extracorporeal bypass. Eur J Cardiothorac Surg. 2009 Aug;36(2):330-4. doi: 10.1016/j.ejcts.2009.03.045. Epub 2009 May 2. PMID 19411180
- [Background] Simons AP, Lance MD, Reesink KD, van der Veen FH, Weerwind PW, Maessen JG. Quantitative assessment of cardiac load-responsiveness during extracorporeal life support: case and rationale. J Cardiothorac Surg. 2010 Apr 27;5:30. doi: 10.1186/1749-8090-5-30. PMID 20423482